CLINICAL TRIAL: NCT02138110
Title: The INSPIRE Study: InVivo Study of Probable Benefit of the Neuro-Spinal Scaffold(TM) for Safety and Neurologic Recovery in Subjects With Complete Thoracic AIS A Spinal Cord Injury
Brief Title: The INSPIRE Study: Probable Benefit of the Neuro-Spinal Scaffold for Treatment of AIS A Thoracic Acute Spinal Cord Injury
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Primary Endpoint not met in follow-up study (InVivo-100-105)
Sponsor: InVivo Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: InVivo-100-101
Record Dates: First submitted 2014-05-01; First posted 2014-05-14 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Traumatic Thoracic Acute Spinal Cord Injury
Keywords: Spinal Cord Injury (SCI); Complete (AIS A) Traumatic Acute Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Neuro-Spinal Scaffold (Experimental): Implantation of a Neuro-Spinal Scaffold into the epicenter of the post-irrigation contusion cavity during open spine surgery
  Interventions: Device: Neuro-Spinal Scaffold

INTERVENTIONS:
Device: Neuro-Spinal Scaffold — Implantation of a Neuro-Spinal Scaffold into the epicenter of the post-irrigation contusion cavity during open spine surgery

SUMMARY:
This is an HDE probable benefit, open-label, non- randomized, single-arm, multicenter study to evaluate the safety and probable benefit of the poly(lactic-co-glycolic acid)-b-poly(L-lysine) Scaffold ("Scaffold") in subjects with thoracic AIS A traumatic spinal cord injury at neurological level of injury of T2-T12.

DETAILED DESCRIPTION:
This is an HDE probable benefit, open-label, non-randomized, single-arm, multicenter study to evaluate the safety and probable benefit of the poly(lactic-co-glycolic acid)-b-poly(L-lysine) Scaffold ("Scaffold") in subjects with thoracic AIS A traumatic spinal cord injury at neurological level of injury of T2-T12.

The study will be conducted by qualified Investigators who have been trained on the surgical Scaffold implant procedure in order to enroll subjects in the Primary Endpoint Analysis Set, defined as all subjects with a successful Scaffold implant, no major protocol deviations, and a complete 6-month Primary Endpoint Follow-up Visit. After receiving the Scaffold and following discharge, subjects will participate in a comprehensive rehabilitation program. For the first 24-months after implantation of the Scaffold, Follow-up and Long-term Follow-up assessments will be conducted at either the study site or the rehabilitation center. The Long-term Follow-up annual visits for years 3 through 10 will be conducted over the telephone.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following to be considered eligible:

1. AIS A classification of traumatic spinal cord injury at T2-T12 neurological level of injury confirmed by a qualified medical professional
2. Recent injury (must receive Scaffold within 7 days from injury)
3. Non-penetrating SCI (contusion injury) that is no less than approximately 4 mm in diameter by MRI
4. Requires open spine surgery allowing access to the injured spinal cord (subjects requiring either posterior surgical approach or posterior plus anterior approach will be eligible)
5. Informed consent obtained
6. 16-70 years of age, inclusive
7. Hemodynamically stable and deemed a suitable candidate for surgery

Exclusion Criteria:

Subjects who meet any of the following will be excluded:

1. Terminally ill subjects not likely to be able to participate in follow-up
2. Incomplete spinal cord injury (AIS B, C, D, and E injuries)
3. Subjects with more than one discrete spinal cord injury (contusion) will be excluded.
4. No discrete cavity (existing or created by irrigation/myelotomy) in the contused spinal cord in which a Scaffold can be placed
5. Evidence of clear and significant Somatosensory Evoked Potentials (SSEP) transmission through the injury site before Scaffold implantation (based on the judgment of the Investigator)
6. Subjects with clinically significant pre-existing neurological comorbidities that are unrelated to the contusion being treated (e.g., multiple sclerosis, amyotrophic lateral sclerosis, significant prior peripheral nerve dysfunction, residual problems related to previous spine-related neurological pathologies) will be excluded only if it is felt that these preexisting morbidities will increase risk, affect safety monitoring, or confound study results
7. Spinal cord injury associated with significant traumatic brain injury or coma that, in the opinion of the Investigator, would preclude adequate assessment of spinal cord function, brain injury that could be associated on its own with sensory or motor deficits, or subjects with any other reason that results in an unreliable International Standards of Neurological Classification of Spinal Cord Injury (ISNCSCI) exam
8. Subjects with clinically significant pre-existing respiratory disease not related to the contusion being treated (e.g., chronic obstructive pulmonary disorder)
9. Subjects requiring Long-term ongoing mechanical ventilation
10. Subjects with documented immune deficiency disorders, including a known diagnosis of HIV infection/AIDS
11. Recent (according to Diagnostic and Statistical Manual of Mental Disorders (DSM) IV or DSM V criteria) history of abuse of narcotics or other significant substance abuse
12. Significant injury complications where, in the view of the Investigator, participation in the study could further complicate subject care, limit study follow-up, or confound interpretation of safety or efficacy data.
13. A female who is:

    * Pregnant, or planning to become pregnant within the next 12-months; or
    * Breastfeeding; or
    * A woman of child-bearing potential (defined as post menarche and biologically capable of becoming pregnant [i.e., not surgically sterile]) who is engaged in active heterosexual relations and is not willing to use a barrier or hormonal form of birth control for 12-months following Scaffold implantation (e.g., oral, injected, or implanted contraceptives)
14. A male who is engaged in active heterosexual relations and is not willing to use birth control for 3-months following Scaffold implantation including sperm donation or banking
15. Current or impending incarceration
16. Complete spinal cord transection
17. Subjects with spinal cord injuries directly due to gunshot, knife, or other penetrating wounds.
18. Known hypersensitivity to poly(lactic-co-glycolic acid) (PLGA) or poly-L-lysine (PLL) (e.g., hypersensitivity to absorbable sutures containing PLGA)
19. History of severe mental illness (according to DSM IV or V)
20. Evidence of pre-trauma active local or systemic infection
21. Participation in another interventional clinical trial for six months after Scaffold implantation
22. Body mass index (BMI) over 39
23. Having a medical condition (e.g., cardiovascular disease, life threatening injuries), or receiving medical treatment, or having any other reason that, in the judgment of the Investigator, precludes successful participation and follow-up for at least six months or confounds collection or interpretation of study safety, feasibility, or efficacy data

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2023-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Toselli, MD, Study Director — InVivo Therapeutics Corporation
Locations (8):
- United States (8):
  - Barrow Neurological Institute - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - USC/Keck School of Medicine, Los Angeles, California
  - University of California/Davis Medical Center, Sacramento, California
  - Cooper Neurological Institute, Camden, New Jersey
  - Carolina NeuroSurgery and Spine Associates/Carolinas Rehabilitation, Charlotte, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Oregon Health & Science University, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harrop JS, Kim KD, Okonkwo DO, Goldstein IM, Lee KS, Toselli RM. Acute Implantation of a Bioresorbable Polymer Scaffold in Patients With Complete Thoracic Spinal Cord Injury: A Randomized Controlled Trial (INSPIRE 2.0). Neurosurgery. 2025 Apr 1;96(4):751-762. doi: 10.1227/neu.0000000000003180. Epub 2024 Oct 8. PMID 39471088
- [Derived] Kim KD, Lee KS, Coric D, Harrop JS, Theodore N, Toselli RM. Acute Implantation of a Bioresorbable Polymer Scaffold in Patients With Complete Thoracic Spinal Cord Injury: 24-Month Follow-up From the INSPIRE Study. Neurosurgery. 2022 Jun 1;90(6):668-675. doi: 10.1227/neu.0000000000001932. Epub 2022 Apr 22. PMID 35442254
- [Derived] Kim KD, Lee KS, Coric D, Chang JJ, Harrop JS, Theodore N, Toselli RM. A study of probable benefit of a bioresorbable polymer scaffold for safety and neurological recovery in patients with complete thoracic spinal cord injury: 6-month results from the INSPIRE study. J Neurosurg Spine. 2021 Feb 5;34(5):808-817. doi: 10.3171/2020.8.SPINE191507. Print 2021 May 1. PMID 33545674
- [Derived] Theodore N, Hlubek R, Danielson J, Neff K, Vaickus L, Ulich TR, Ropper AE. First Human Implantation of a Bioresorbable Polymer Scaffold for Acute Traumatic Spinal Cord Injury: A Clinical Pilot Study for Safety and Feasibility. Neurosurgery. 2016 Aug;79(2):E305-12. doi: 10.1227/NEU.0000000000001283. PMID 27309344

RESULTS

PARTICIPANT FLOW:
Period: Enrolled in Study
Arm/Group | Neuro-Spinal Scaffold
Started | 20
Completed | 20
Not Completed | 0
Period: Enrolled for Scaffold Implantation
Arm/Group | Neuro-Spinal Scaffold
Started | 20
Completed | 19
Not Completed | 1
Not completed — Physician Decision | 1
Period: Overall Scaffold Implantation
Arm/Group | Neuro-Spinal Scaffold
Started | 19
6-month Follow-Up | 16
Completed | 16
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Population: All enrolled subjects minus screen failures.
Groups:
- Neuro-Spinal Scaffold: Implantation of neuro-spinal scaffold in a cavity at the epicenter of the spinal cord contusion during open spine surgery.
  Neuro-Spinal Scaffold
Arm/Group | Neuro-Spinal Scaffold
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: years] | 36 [18 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 1
  Race: Black or African American | 2
  Race: White | 16
  Race: Other | 1
Height [Mean (Full Range); unit: cm] | 172 [147 to 185]
Weight [Mean (Full Range); unit: kg] | 83 [58 to 127]
Body Mass Index [Mean (Full Range); unit: kg/m^2] | 28 [20 to 38]
Cause of Injury [Count of Participants; unit: Participants]
  Fall | 5
  Other-All Terrain Vehicle | 1
  Vehicular | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Improvement in AIS Grade of One or More Levels
Description: The ASIA (American Spinal Injury Association) Impairment Scale (AIS) classifies spinal cord injuries as follows:
  A = Complete: no sensory or motor function is preserved in the sacral segments S4-S5
  B = Sensory incomplete: sensory but not motor function is preserved below the neurological level and includes the sacral segments S4-S5, AND no motor function is preserved more than three levels below the motor level on either side of the body
  C = Motor incomplete: motor function is preserved below the neurological level, and more than half of key muscle functions below the single neurological level of injury have a muscle grade less than 3 (Grades 0-2)
  D = Motor incomplete: at least half (half or more) of key muscle functions below the NLI have a muscle grade >3
  E = Normal
  The confirmatory ISNCSCI exam performed within 8 hours prior to surgery was used as the baseline visit.
Time Frame: 6 months post-implantation
Population: The Primary Endpoint Analysis Set includes all subjects who had a successful Neuro-Spinal Scaffold implant, no major data protocol deviations, and completed the 6-month Primary Endpoint Follow-up Visit.
Measure: Number; unit: percentage of patients
Arm/Group | Neuro-Spinal Scaffold
Number analyzed (Participants) | 16
percentage of patients | 44

2. Secondary Outcome: Number of Participants Stratified by Change From Baseline in Neurological Level of Injury (NLI) at 6 Months
Description: The neurological level of injury (NLI) refers to the most caudal segment of the spinal cord with normal sensory and antigravity motor function on both sides of the body, provided that there is normal (intact) sensory and motor function rostrally.
  A caudal change is an improvement in NLI whereas a rostral change is a deterioration in NLI.
  The confirmatory ISNCSCI exam performed within 8 hours prior to surgery was used as the baseline visit.
Time Frame: 6 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Neuro-Spinal Scaffold
Number analyzed (Participants) | 16
Participants
  Caudal change in NLI from baseline | 5
  Rostral change in NLI from baseline | 8
  No change in NLI from baseline | 3

3. Secondary Outcome: Number of Participants Stratified by Change From Baseline in ISNCSCI Sensory Pin Prick Score
Description: International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Sensory Pin Prick Scores were assessed on a scale from 0 to 2 for each sensory point tested on each side of the body (maximum score = 112), with higher scores indicating better neurologic function.
  The confirmatory ISNCSCI exam performed within 8 hours prior to surgery was used as the baseline visit.
  An improvement in pin prick score indicates an increase in score from baseline at 6-months A deterioration in pin prick score indicates a decrease in score from baseline at 6-months No change in pin prick score indicates no change in score from baseline at 6-months
Time Frame: 6 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Neuro-Spinal Scaffold
Number analyzed (Participants) | 16
Participants
  Improvement | 10
  Deterioration | 6
  No change | 0

4. Secondary Outcome: Number of Participants Stratified by Change From Baseline in ISNCSCI Sensory Light Touch Score
Description: International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Sensory Light Touch Scores were assessed on a scale from 0 to 2 for each sensory point tested on each side of the body (maximum score = 112), with higher scores indicating better neurologic function.
  The confirmatory ISNCSCI exam performed within 8 hours prior to surgery was used as the baseline visit.
  An improvement in light touch score indicates an increase in light touch score from baseline at 6-months A deterioration in light touch score indicates a decrease in light touch score from baseline at 6-months No change in light touch score indicates no change in light touch score from baseline at 6-months
Time Frame: 6 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Neuro-Spinal Scaffold
Number analyzed (Participants) | 16
Participants
  Improvement | 10
  Deterioration | 4
  No change | 2

5. Secondary Outcome: Change From Baseline in ISNCSCI Total Motor Score
Description: International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) Total Motor Scores were assessed on a scale from 0 to 5 for each myotome tested on each side of the body (upper limb maximum score = 50 and lower limb maximum score = 50), with higher scores indicating better neurologic function.
  The confirmatory ISNCSCI exam performed within 8 hours prior to surgery was used as the baseline visit.
  An improvement in motor score indicates an increase in motor score from baseline at 6-months A deterioration in motor score indicates an decrease in motor score from baseline at 6-months No change in motor score indicates no change in motor score from baseline at 6-months
Time Frame: 6 months post-implantation
Population: Results from 15 of 16 patients are presented. This is because pre-implantation assessment was not testable for 1 of 16 patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Neuro-Spinal Scaffold
Number analyzed (Participants) | 15
Participants
  Improvement | 1
  Deterioration | 0
  No Change | 14

6. Secondary Outcome: Number of Participants Stratified by Change From Baseline in Spinal Cord Anatomy - Cyst (Presence or Absence)
Description: Characteristics of spinal cord anatomy were assessed by a Board-certified neuroradiologist central reader including presence or absence of intraparenchymal cysts.
  Screening MRI was used as the baseline value.
Time Frame: 6 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Neuro-Spinal Scaffold
Number analyzed (Participants) | 16
Participants
  Cyst Detected | 9
  No Cyst Detected | 5
  Indeterminate | 2

7. Secondary Outcome: Number of Participants Stratified by Change From Baseline in Spinal Cord Anatomy - Spinal Cord Adhesion (Presence or Absence)
Description: Characteristics of spinal cord anatomy were assessed by a Board-certified neuroradiologist central reader including the presence or absence of spinal cord adhesion.
  Screening MRI was used as the baseline value.
Time Frame: 6 months post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Neuro-Spinal Scaffold
Number analyzed (Participants) | 16
Participants
  Spinal Cord Adhesion Detected | 1
  No Spinal Cord Adhesion Detected | 13
  Indeterminate | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the implantation of scaffold through the 6 month primary endpoint follow-up visit from to the 12 month follow-up for the subjects that reached this time point at the time of analysis.
Arm/Group | Neuro-Spinal Scaffold
All-Cause Mortality (participants affected / at risk) | 3/19
Serious Adverse Events (participants affected / at risk) | 19/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuro-Spinal Scaffold (N=19)
Colitis (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (4)
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Necrotising myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Spinal cord disorder (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuro-Spinal Scaffold (N=19)
Anaemia (Blood and lymphatic system disorders) | 3 (4)
Leukocytosis (Blood and lymphatic system disorders) | 6 (7)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 6 (6)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Anal fissure (Gastrointestinal disorders) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 3 (4)
Dry mouth (Gastrointestinal disorders) | 2 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (5)
Proctitis (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Tooth impacted (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Adverse drug reaction (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Generalised oedema (General disorders) | 1 (1)
Medical device complication (General disorders) | 1 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Pyrexia (General disorders) | 8 (8)
Systemic inflammatory response syndrome (General disorders) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Candiduria (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Cellulitis of male external genital organ (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Enterococcal infection (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Serratia infection (Infections and infestations) | 1 (1)
Streptococcal urinary tract infection (Infections and infestations) | 1 (1)
Tinea pedis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 12 (38)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1)
Chemical peritonitis (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (2)
Incision site pain (Injury, poisoning and procedural complications) | 4 (4)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Nail avulsion (Injury, poisoning and procedural complications) | 1 (1)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 2 (3)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Ammonia increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (2)
Blood creatinine increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blood prolactin increased (Investigations) | 1 (1)
Blood urea increased (Investigations) | 1 (1)
Body temperature fluctuation (Investigations) | 1 (1)
Body temperature increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Hepatic enzyme increased (Investigations) | 1 (1)
Red blood cell sedimentation rate increased (Investigations) | 1 (1)
White blood cell count increased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (4)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (15)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Necrotising myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (9)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Syringomyelia (Nervous system disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysaesthesia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (5)
Lethargy (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 2 (2)
Muscle spasticity (Nervous system disorders) | 4 (6)
Myelomalacia (Nervous system disorders) | 2 (3)
Neuralgia (Nervous system disorders) | 10 (12)
Neurological decompensation (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Poor quality sleep (Nervous system disorders) | 1 (1)
Spinal meningeal cyst (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Acute stress disorder (Psychiatric disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (4)
Depression (Psychiatric disorders) | 5 (8)
Insomnia (Psychiatric disorders) | 3 (3)
Mood swings (Psychiatric disorders) | 1 (1)
Bladder pain (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Incontinence (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 4 (4)
Acquired hydrocele (Reproductive system and breast disorders) | 2 (2)
Galactorrhoea (Reproductive system and breast disorders) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 1 (1)
Scrotal oedema (Reproductive system and breast disorders) | 1 (1)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 2 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 5 (7)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 3 (4)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1)
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
Hypotension (Vascular disorders) | 4 (4)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1)
Venous occlusion (Vascular disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 1 (1)
Injection site pain (General disorders) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Autonomic dysreflexia (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-06-29): https://cdn.clinicaltrials.gov/large-docs/10/NCT02138110/Prot_002.pdf
  • Statistical Analysis Plan (2018-01-17): https://cdn.clinicaltrials.gov/large-docs/10/NCT02138110/SAP_000.pdf